CLINICAL TRIAL: NCT03714789
Title: Clearance and Pharmacokinetics of Antibiotics With Different Protein-bound Levels in Renal Replacement Therapy
Brief Title: Clearance and Pharmacokinetics of Antibiotics in Renal Replacement Therapy
Status: Completed | Type: Observational
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Collaborators: Institute of Antibiotics, Huashan Hospital, Fudan University (Unknown)
Responsible Party: Principal Investigator, Ding Feng, Kidney internal medicine professor, Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Other Study IDs: PKDialysis-201710
Record Dates: First submitted 2018-10-14; First posted 2018-10-22 (Actual); Last update posted 2020-10-26 (Actual); Status verified 2020-10

CONDITIONS: Kidney Failure
Keywords: Kidney Failure; Pharmacokinetics; Antibiotics
MeSH Terms: conditions — Renal Insufficiency | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Meropenem: Patients requiring dialysis and receiving meropenem for infection or suspended infection.
  Interventions: Other: Blood and spent dialysate collection
- Vancomycin: Patients requiring dialysis and receiving vancomycin for infection or suspended infection.
  Interventions: Other: Blood and spent dialysate collection
- Ceftriaxone: Patients requiring dialysis and receiving ceftriaxone for infection or suspended infection.
  Interventions: Other: Blood and spent dialysate collection

INTERVENTIONS:
Other: Blood and spent dialysate collection — A certain amount of blood and spent dialysate are collected during and after dialysis for quantification of drug concentration.

SUMMARY:
This is an observational study that evaluates the dialysis clearance and pharmacokinetics of antibiotics with different protein-bound levels in patients receiving renal replacement therapy. Meropenem, vancomycin and ceftriaxone are selected to represent three typical protein-bound levels, and the primary dialysis methods being studied are intermittent hemodialysis(IHD) and hemodiafiltration(HDF). During and after the dialysis, the drug levels in both plasma and spent dialysate are monitored, but no changes are made to therapy. The study will provide detailed information on the characteristics of the removal kinetics of the three antibiotics during dialysis, and evaluate whether the dosing regimens are the most appropriate to achieve therapeutic targets while minimizing the risk of toxicity.

DETAILED DESCRIPTION:
This prospective, single-center observational study is taken to evaluate the dialysis clearance and pharmacokinetics of antibiotics with three different protein-bound levels in patients receiving renal replacement therapy. As is known that the plasma protein binding rate affects the distribution, metabolism and elimination of the drug in the body, and is also an important factor affecting the removal during dialysis, the study selects meropenem, vancomycin and ceftriaxone, of which the protein-bound levels are respectively 2%, 55% and 85%, to represent three typical protein-bound levels. The primary dialysis methods being studied are intermittent hemodialysis(IHD) and hemodiafiltration(HDF). The dialysis pattern, the antibiotic choice and its dosage for each subject are made on clinical grounds. A total of 16 milliliters of blood and 60 milliliters of spent dialysate are collected from each subject for each dialysis pattern. The study will provide detailed information on the characteristics of the removal kinetics of the three antibiotics during dialysis, and evaluate whether the dosing regimens are the most appropriate to achieve therapeutic targets while minimizing the risk of toxicity.

ELIGIBILITY:
Inclusion Criteria:

* With Age from 18 to 85 years old.
* With weight from 50 to 75 kilograms.
* Requiring dialysis including intermittent hemodialysis(IHD) or hemodiafiltration(HDF).
* Receiving meropenem, vancomycin or ceftriaxone based on clinical grounds.

Exclusion Criteria:

* Patient is during pregnant or lactation period.
* Patient is allergic to meropenem, vancomycin or ceftriaxone.
* Severe hypoproteinemia (serum total protein<=45g/L) or severe hypoalbuminemia（serum albumin<20g/L).
* Severe liver dysfunction（ALT>200U/L or AST>200U/L).
* The patient himself or his immediate family refuses to sign the informed consent.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients aged from 18 to 85 years, requiring dialysis including intermittent hemodialysis(IHD) or hemodiafiltration(HDF), and receiving meropenem, vancomycin or ceftriaxone based on clinical grounds from a university-affiliated hospital in Shanghai, China.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Dialytic clearance (K_total) | During the session of dialysis, up to 4 hours
  The total drug amount removed by dialysis
Area under the concentration-time curve (AUC) | During the session of dialysis, up to 4 hours
  AUC based on plasma concentration during dialysis

SECONDARY OUTCOMES:
Rebound of plasma concentration (Rebound_1h%) | At the end of dialysis and an hour after dialysis
  The rebound rate of plasma concentration 1 hour after dialysis

CONTACTS AND LOCATIONS:
Overall Officials: Feng Ding, PhD, Study Director — Division of Nephrology,Shanghai Ninth People's Hospital, School of Medicine, Shanghai Jiaotong University
Locations (1):
- Shanghai Ninth People's Hospital, Shanghai, China